CLINICAL TRIAL: NCT05243745
Title: An 8-week, Randomised, Controlled, Examiner-Blind, Proof of Principle Study Investigating the Ability of a 3% Methyl Vinyl Ether/Maleic Anhydride Co-Polymer (PVM/MA) + 5% Potassium Nitrate (KNO3) Combination Toothpaste to Protect From Dentine Hypersensitivity
Brief Title: Exploratory Clinical Study to Investigate the Ability of an Experimental Combination Dentifrice to Protect Sensitive Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 218220
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Product (Experimental): Participants will dose the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Test product is a combination toothpaste of 3% methyl vinyl ether/maleic anhydride co-polymer (PVM/MA) + 5% Potassium Nitrate (KNO3). Participants will brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening); Participants will be permitted to rinse with water post-brushing.
  Interventions: Other: 3% PVM/MA + 5% KNO3 Combination
- Comparator 1 (Active Comparator): Participants will dose the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Comparator 1 toothpaste is containing 3% PVM/MA. Participants will brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening); participants will be permitted to rinse with water post-brushing.
  Interventions: Other: 3% PVM/MA only
- Comparator 2 (Active Comparator): Participants will dose the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Comparator 2 toothpaste is containing 5% KNO3. Participants will brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening); participants will be permitted to rinse with water post-brushing.
  Interventions: Other: 5% KNO3 Only
- Negative Control (Other): Participants will dose the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Negative control is regular fluoride toothpaste. Participants will brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening); participants will be permitted to rinse with water post-brushing.
  Interventions: Other: Regular Fluoride

INTERVENTIONS:
Other: 3% PVM/MA + 5% KNO3 Combination — Toothpaste containing 3% PVM/MA + 5% KNO3 as combination will be used as test product.
  Arms: Test Product
Other: 3% PVM/MA only — Toothpaste containing 3% PVM/MA only will be used as comparator 1 product.
  Arms: Comparator 1
Other: 5% KNO3 Only — Toothpastes containing 5% KNO3 only will be used as comparator 2 product.
  Arms: Comparator 2
Other: Regular Fluoride — Toothpaste containing regular fluoride will be used as negative control.
  Arms: Negative Control

SUMMARY:
This proof of principle (PoP) study will evaluate the ability of an experimental combination toothpaste formulation to protect sensitive teeth from dentine hypersensitivity.

DETAILED DESCRIPTION:
This will be a PoP, single centre, 8-week, randomised, controlled, examiner blind, parallel design, stratified (by maximum Baseline Schiff sensitivity score of the two selected test teeth) clinical study in healthy participants with sensitive teeth.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent indicating the participant has been informed of all pertinent aspects of the study before any study procedures are performed.
* Participant who is willing and able to comply with scheduled visits, product usage requirements and other study procedures.
* Participant in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history, or upon oral examination, that would impact the participant's safety or wellbeing, or the outcomes of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Female participant of child-bearing potential and at risk for pregnancy who agrees to use a highly effective method of contraception throughout the study and for at least 5 days after the last use of assigned study product.
* AT VISIT 1 (Screening):

Participant must have

1. a self-reported history of tooth sensitivity lasting more than six months but not more than 10 years.
2. a minimum of 20 natural teeth.
3. a minimum of 2 accessible, non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, with clinically confirmed DH; each tooth must meet the following criteria:

   * exposed dentine due to facial/cervical erosion, abrasion or gingival recession (EAR).
   * MGI score = 0 adjacent to the test area (exposed dentine) only (Lobene et al.,1986)
   * clinical mobility = 0 (Laster et al., 1975)
   * Dentin Hypersensitivity (DH) as evidenced by qualifying levels of tactile and evaporative (air) sensitivity (tactile threshold less than or equal to <= 20 gram (g); Schiff sensitivity score greater than or equal to >= 2).
   * AT VISIT 2 (Baseline):

Participant must have a minimum of two, non-adjacent accessible teeth (incisors, canines, pre molars) with DH, as evidenced by qualifying levels of tactile and evaporative (air) sensitivity (tactile threshold less than or equal to <= 20 g; Schiff sensitivity score >= 2) at the Screening and Baseline visits.

Note: All teeth which meet the eligibility criteria at Screening (Visit 1) should be assessed by tactile and evaporative (air) stimuli at Baseline (Visit 2).

The examiner will select two 'test teeth' from those which meet the tactile threshold and Schiff sensitivity score inclusion criteria at both Screening and Baseline. Test teeth should not be adjacent to each other and preferably in different quadrants.

Exclusion Criteria:

* Participant who is an employee of the study site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the study site otherwise supervised by the investigator; or a GlaxoSmithKline Consumer Healthcare (GSK CH) employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days of study entry and/or during study participation.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Female participant who is pregnant (as evidenced by a positive urine pregnancy test (UPT) at Screening) or intending to become pregnant during the study.
* Female participant who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to the study products or any of their stated ingredients (or closely related compounds).
* Participant who is unwilling or unable to comply with the Lifestyle Considerations.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* Participant who has participated in another tooth sensitivity study within 8 weeks of Screening.
* Participant who has used an oral care product indicated for the relief of DH or care of sensitive teeth within 8 weeks of Screening (participants will be required to verbally confirm the name of their current oral care products to enable site staff to verify the absence of known sensitivity ingredients).
* Participant who has had dental prophylaxis within 4 weeks of Screening.
* Participant who has had a teeth bleaching procedure within 8 weeks of Screening.
* Participant who has had treatment for periodontal disease (including surgery) within 12 months of Screening.
* Participant who has had scaling or root planning within 3 months of Screening.
* Participant with gross periodontal disease.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with a tongue or lip piercing.
* Participant with a fixed or removable partial prosthesis which, in the opinion of the investigator, would impact study outcomes.
* Participant with multiple dental implants which, in the opinion of the investigator, would impact study outcomes.
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* SPECIFIC DENTITION EXCLUSIONS FOR 'TEST TEETH':

  1. Tooth with evidence of current or recent caries or reported treatment of decay within 12 months of Screening.
  2. Tooth with exposed dentine but with deep, defective or facial restorations.
  3. Tooth with full crown or veneer.
  4. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator, would impact study outcomes.
  5. Sensitive tooth with contributing etiologies other than erosion, abrasion or recession to exposed dentine.
  6. Sensitive tooth not expected to benefit from use of a sensitivity toothpaste in the opinion of the investigator
* Participant taking daily doses of medication/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, antidepressants, mood-altering and anti-inflammatory drugs).
* AT VISIT 1 (Screening):

Participant who has taken antibiotics in the 2 weeks prior to the Screening visit.

- AT VISIT 2 (Baseline): Participant who has taken antibiotics in the 2 weeks prior to the Baseline visit, during the acclimatisation period.

* Participant who is taking daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant who requires antibiotic prophylaxis for dental procedures.
* Participant who has previously been enrolled in this study.
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Dental School, University of Bristol, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 133 participants were screened of which 120 participants were randomized to a treatment with either one of the 4 products: test product (combination toothpaste of 3 percent [%] methyl vinyl ether/maleic anhydride co-polymer [PVM/MA] + 5% Potassium Nitrate [KNO3]), comparator 1 (toothpaste containing 3% PVM/MA), comparator 2 (toothpaste containing 5% KNO3), or negative control (a regular fluoride toothpaste).
Groups:
- Test Product: Participants were dosed by the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Test product was a combination toothpaste of 3 % PVM/MA + 5% KNO3. Participants were instructed to brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening) for 8 weeks. Participants were permitted to rinse with water post-brushing.
- Comparator 1: Participants were dosed by the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Comparator 1 was a toothpaste containing 3% PVM/MA. Participants were instructed to brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening) for 8 weeks. Participants were permitted to rinse with water post-brushing.
- Comparator 2: Participants were dosed by the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Comparator 2 was a toothpaste containing 5% KNO3. Participants were instructed to brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening) for 8 weeks. Participants were permitted to rinse with water post-brushing.
- Negative Control: Participants were dosed by the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Negative control was a regular fluoride toothpaste. Participants were instructed to brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening) for 8 weeks. Participants were permitted to rinse with water post-brushing.
Period: Overall Study
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Started | 29 | 31 | 31 | 29
Completed | 29 | 31 | 30 | 28
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Unable to Attend Visit 6 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who completed at least one use of study product.
Groups:
- Test Product: Participants were dosed by the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion. Test product was a combination toothpaste of 3% PVM/MA + 5% KNO3. Participants were instructed to brush their two selected 'test teeth' first, followed by the whole mouth for one timed minute, twice daily (morning and evening) for 8 weeks. Participants were permitted to rinse with water post-brushing.
- Total: Total of all reporting groups
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control | Total
Number analyzed (Participants) | 29 | 31 | 31 | 29 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.93) | 41.5 (12.20) | 41.9 (14.29) | 40.9 (15.10) | 42.2 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 25 | 26 | 22 | 91
  Male | 11 | 6 | 5 | 7 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 1 | 0 | 4 | 6
  Asian - Central/South Asian Heritage | 3 | 1 | 3 | 1 | 8
  Asian - South East Asian Heritage | 0 | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 25 | 29 | 26 | 24 | 104
  Multiple | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Baseline (Day 0)
Description: Evaporative (air) sensitivity was assessed on facial surfaces of eligible incisor,canine and pre-molar teeth by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface,approximately 1-2 millimeter(mm) coronal to gingival margin from a distance of approximately 1 centimeter(cm). Participant response to the stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative stimulus. Score ranged from 0-3; 0=Did not respond to air stimulation;1=Responded to air stimulus but did not request discontinuation of stimulus;2=Responded to air stimulus and requested discontinuation or moved from stimulus;3=Responded to stimulus, considered stimulus to be painful, requested discontinuation of stimulus. A decrease in Schiff sensitivity score indicated an improvement in sensitivity. Mean was calculated once by selecting 2 test teeth located in different quadrants of mouth.
Time Frame: Baseline (Day 0)
Population: The modified intent-to-treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one post-baseline clinical performance assessment (Schiff sensitivity assessment or Tactile sensitivity assessment).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale | 2.43 (0.438) | 2.44 (0.442) | 2.44 (0.442) | 2.34 (0.356)

2. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 3
Description: Evaporative (air) sensitivity was assessed on facial surfaces of eligible incisor, canine and pre-molar teeth by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface, approximately 1-2 mm coronal to gingival margin from a distance of approximately 1 cm. Participant response to the stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative stimulus. Score ranged from 0-3; 0=Did not respond to air stimulation;1=Responded to air stimulus but did not request discontinuation of stimulus;2=Responded to air stimulus and requested discontinuation or moved from stimulus;3=Responded to stimulus, considered stimulus to be painful, requested discontinuation of stimulus. A decrease in Schiff sensitivity score indicated an improvement in sensitivity. Mean was calculated once by selecting 2 test teeth located in different quadrants of mouth.
Time Frame: Day 3
Population: The mITT population. Here, overall number analyzed is the number of participants with data available for analyses for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 28 | 29 | 28
score on a scale | 1.31 (0.618) | 1.41 (0.681) | 1.88 (0.456) | 2.09 (0.431)

3. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 14
Description: as for outcome 2
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 27 | 29 | 30 | 29
score on a scale | 0.69 (0.419) | 1.00 (0.567) | 1.37 (0.414) | 2.10 (0.387)

4. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 28
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 25 | 30 | 30 | 26
score on a scale | 0.52 (0.510) | 0.92 (0.588) | 1.13 (0.414) | 2.10 (0.375)

5. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 56
Description: as for outcome 2
Time Frame: Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 30 | 28
score on a scale | 0.33 (0.449) | 0.69 (0.441) | 1.17 (0.547) | 2.02 (0.396)

6. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Baseline (Day 0)
Description: Tactile sensitivity was assessed for eligible incisor, canine and pre-molar teeth using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting at which participant gave two consecutive 'yes' responses was recorded as the tactile threshold (grams [g]). At Baseline, the maximum force was 20 g; at all subsequent visits, 80 g. If no sensitivity was found at the upper limit, the tactile threshold was recorded as greater than (>) 20 g (baseline) or >80 g (all other visits). An increase in tactile threshold indicated an improvement. Mean was calculated once by selecting two test teeth which were located in different quadrants of mouth.
Time Frame: Baseline (Day 0)
Population: The mITT population.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
grams | 12.76 (3.429) | 11.94 (3.577) | 12.74 (4.049) | 12.24 (3.681)

7. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 3
Description: Tactile sensitivity was assessed for eligible incisor, canine and pre-molar teeth using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting at which participant gave two consecutive 'yes' responses was recorded as the tactile threshold (g). At Baseline, the maximum force was 20 g; at all subsequent visits, 80 g. If no sensitivity was found at the upper limit, the tactile threshold was recorded as >20 g (baseline) or >80 g (all other visits). An increase in tactile threshold indicated an improvement. Mean was calculated once by selecting two test teeth which were located in different quadrants of mouth.
Time Frame: Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 28 | 29 | 28
grams | 46.38 (12.528) | 40.00 (9.718) | 27.59 (9.026) | 22.14 (7.985)

8. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 14
Description: as for outcome 7
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 27 | 29 | 30 | 29
grams | 58.15 (11.107) | 48.62 (8.752) | 40.33 (8.087) | 24.83 (7.498)

9. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 28
Description: as for outcome 7
Time Frame: Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 25 | 30 | 30 | 26
grams | 62.60 (12.675) | 51.83 (9.237) | 48.50 (8.320) | 25.38 (5.463)

10. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 56
Description: as for outcome 7
Time Frame: Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 30 | 28
grams | 67.93 (12.992) | 58.23 (11.514) | 48.83 (9.886) | 28.57 (6.920)

11. Primary Outcome: Mean Number of Sensitive Teeth (Schiff Sensitivity Score Greater Than or Equal to [>=] 1) at Baseline (Day 0)
Description: Sensitive teeth were defined as teeth with Schiff sensitivity score of >=1 (Schiff sensitivity scale: 0=Participant did not respond to air stimulation; 1=Participant responded to air stimulus but did not request discontinuation of stimulus; 2=Participant responded to air stimulus and requested discontinuation or moved from stimulus; 3=Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus). A decrease in the mean number of sensitive teeth indicated an improvement in sensitivity.
Time Frame: Baseline (Day 0)
Population: The mITT population.
Measure: Mean (Standard Deviation); unit: sensitive teeth
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
sensitive teeth | 3.79 (1.373) | 3.68 (1.137) | 3.68 (1.249) | 3.24 (0.577)

12. Primary Outcome: Mean Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 3
Description: as for outcome 11
Time Frame: Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: sensitive teeth
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 28 | 29 | 28
sensitive teeth | 3.48 (1.573) | 3.36 (1.367) | 3.72 (1.279) | 3.25 (0.585)

13. Primary Outcome: Mean Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 14
Description: as for outcome 11
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: sensitive teeth
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 27 | 29 | 30 | 29
sensitive teeth | 2.59 (1.394) | 3.10 (1.496) | 3.60 (1.303) | 3.24 (0.577)

14. Primary Outcome: Mean Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 28
Description: as for outcome 11
Time Frame: Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: sensitive teeth
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 25 | 30 | 30 | 26
sensitive teeth | 2.24 (2.026) | 2.93 (1.617) | 3.30 (1.466) | 3.27 (0.604)

15. Primary Outcome: Mean Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 56
Description: as for outcome 11
Time Frame: Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: sensitive teeth
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 30 | 28
sensitive teeth | 1.72 (1.771) | 2.35 (1.380) | 3.17 (1.621) | 3.25 (0.585)

16. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Days 3, 14, 28 and 56
Description: Evaporative (air) sensitivity was assessed on facial surfaces of teeth by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface,approximately 1-2 mm coronal to gingival margin from approximately 1 cm. Participant response to stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative stimulus. Score ranged from 0-3;0=Did not respond to air stimulation;1=Responded to air stimulus but did not request discontinuation of stimulus;2=Responded to air stimulus and requested discontinuation or moved from stimulus;3=Responded to stimulus, considered stimulus to be painful, requested discontinuation of stimulus. A decrease in Schiff sensitivity score indicated an improvement in sensitivity. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A negative change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 2.43 (0.438) | 2.44 (0.442) | 2.44 (0.442) | 2.34 (0.356)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | -1.12 (0.622) | -1.04 (0.666) | -0.57 (0.513) | -0.25 (0.347)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | -1.70 (0.505) | -1.43 (0.513) | -1.05 (0.531) | -0.24 (0.344)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -1.94 (0.441) | -1.53 (0.556) | -1.32 (0.445) | -0.29 (0.404)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -2.10 (0.507) | -1.74 (0.546) | -1.28 (0.552) | -0.34 (0.361)
Statistical Analysis 1: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 3; Test type: Superiority; p = 0.4990, ANCOVA; Analysis was performed using ANCOVA model with study product as a factor and baseline Schiff sensitivity score as a covariate; Adjusted Mean Difference = -0.09, 95% CI 2-sided [-0.36 to 0.18], Standard Error of Mean 0.136 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 2: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 3; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.56, 95% CI 2-sided [-0.83 to -0.29], Standard Error of Mean 0.135 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 3: Comparison: Test Product vs Negative Control; Change from Baseline at Day 3; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.83, 95% CI 2-sided [-1.10 to -0.56], Standard Error of Mean 0.137 — Adjusted Mean Difference is calculated as Test value minus Negative Control value
Statistical Analysis 4: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 14; Test type: Superiority; p = 0.0090, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.30, 95% CI 2-sided [-0.52 to -0.08], Standard Error of Mean 0.112 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 5: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 14; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.67, 95% CI 2-sided [-0.89 to -0.45], Standard Error of Mean 0.111 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 6: Comparison: Test Product vs Negative Control; Change from Baseline at Day 14; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -1.44, 95% CI 2-sided [-1.66 to -1.22], Standard Error of Mean 0.112 — Adjusted Mean Difference was calculated as Test value minus Negative Control value
Statistical Analysis 7: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 28; Test type: Superiority; p = 0.0007, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.40, 95% CI 2-sided [-0.63 to -0.17], Standard Error of Mean 0.116 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 8: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.62, 95% CI 2-sided [-0.85 to -0.39], Standard Error of Mean 0.116 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 9: Comparison: Test Product vs Negative Control; Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -1.62, 95% CI 2-sided [-1.85 to -1.38], Standard Error of Mean 0.120 — Adjusted Mean Difference was calculated as Test value minus Negative Control value
Statistical Analysis 10: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 56; Test type: Superiority; p = 0.0015, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.36, 95% CI 2-sided [-0.59 to -0.14], Standard Error of Mean 0.112 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 11: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 56; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -0.83, 95% CI 2-sided [-1.05 to -0.61], Standard Error of Mean 0.113 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 12: Comparison: Test Product vs Negative Control; Change from Baseline at Day 56; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Adjusted Mean Difference = -1.72, 95% CI 2-sided [-1.95 to -1.49], Standard Error of Mean 0.115 — Adjusted Mean Difference was calculated as Test value minus Negative Control

17. Secondary Outcome: Change From Baseline in Tactile Threshold at Days 3, 14, 28 and 56
Description: Tactile sensitivity was assessed for teeth using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting at which participant gave two consecutive 'yes' responses was recorded as the tactile threshold (g). At Baseline, the maximum force was 20 g; at all subsequent visits, 80 g. If no sensitivity was found at the upper limit, the tactile threshold was recorded as >20 g (baseline) or >80 g (all other visits). An increase in tactile threshold indicated an improvement. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A positive change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
grams
  Baseline (Day 0) | 12.76 (3.429) | 11.94 (3.577) | 12.74 (4.049) | 12.24 (3.681)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | 33.62 (11.642) | 27.86 (10.131) | 15.34 (7.898) | 9.82 (8.442)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | 45.19 (9.556) | 36.55 (8.462) | 27.50 (8.279) | 12.59 (7.975)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | 49.60 (12.493) | 40.17 (9.421) | 36.00 (7.812) | 13.85 (5.883)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | 55.17 (12.711) | 46.29 (12.448) | 36.00 (10.372) | 16.61 (8.057)
Statistical Analysis 1: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 3; Test type: Superiority; p = 0.0231, ANCOVA; Analysis was performed using ANCOVA model with study product, baseline Schiff stratification as a factor and baseline tactile threshold as covariate; Adjusted Mean Difference = 5.93, 95% CI 2-sided [0.83 to 11.02], Standard Error of Mean 2.572 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 2: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 3; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 18.42, 95% CI 2-sided [13.37 to 23.47], Standard Error of Mean 2.549 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 3: Comparison: Test Product vs Negative Control; Change from Baseline at Day 3; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 23.93, 95% CI 2-sided [18.83 to 29.02], Standard Error of Mean 2.571 — Adjusted Mean Difference was calculated as Test value minus Negative Control
Statistical Analysis 4: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 14; Test type: Superiority; p = 0.0002, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 8.97, 95% CI 2-sided [4.43 to 13.51], Standard Error of Mean 2.293 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 5: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 14; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Slope = 17.71, 95% CI 2-sided [13.22 to 22.20], Standard Error of Mean 2.265 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 6: Comparison: Test Product vs Negative Control; Change from Baseline at Day 14; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 32.81, 95% CI 2-sided [28.27 to 37.34], Standard Error of Mean 2.288 — Adjusted Mean Difference was calculated as Test value minus Negative Control
Statistical Analysis 7: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 10.20, 95% CI 2-sided [5.28 to 15.13], Standard Error of Mean 2.485 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 8: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 13.92, 95% CI 2-sided [9.05 to 18.80], Standard Error of Mean 2.460 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 9: Comparison: Test Product vs Negative Control; Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 36.51, 95% CI 2-sided [31.42 to 41.60], Standard Error of Mean 2.568 — Adjusted Mean Difference was calculated as Test value minus Negative Control
Statistical Analysis 10: Comparison: Test Product vs Comparator 1; Change from Baseline at Day 56; Test type: Superiority; p = 0.0006, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 9.73, 95% CI 2-sided [4.26 to 15.20], Standard Error of Mean 2.761 — Adjusted Mean Difference was calculated as Test value minus Comparator 1 value
Statistical Analysis 11: Comparison: Test Product vs Comparator 2; Change from Baseline at Day 56; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 19.06, 95% CI 2-sided [13.57 to 24.55], Standard Error of Mean 2.772 — Adjusted Mean Difference was calculated as Test value minus Comparator 2 value
Statistical Analysis 12: Comparison: Test Product vs Negative Control; Change from Baseline at Day 56; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 17, analysis 1]; Adjusted Mean Difference = 39.33, 95% CI 2-sided [33.73 to 44.94], Standard Error of Mean 2.829 — Adjusted Mean Difference was calculated as Test value minus Negative Control value

18. Secondary Outcome: Change From Baseline in Mean Score of Dentine Hypersensitivity Experience Questionnaire (DHEQ) (Section 1 Questions 7-9) at Days 3, 14, 28 and 56
Description: The DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of two sections. Section 1 included 9 questions about participant's sensitive teeth and the impact it has on participant's everyday life. All participants scored question number 7 to 9. Question (Q)7 (On a scale of 1 to 10 how intense are the sensations) was scored from 1=not at all intense to 10=worst imaginable; Q8 (On a scale of 1 to 10 how bothered are you by any sensations?) was scored from 1=not at all bothered to 10=extremely bothered; Q9 (On a scale of 1 to 10 how well you can tolerate the sensations?) was scored from 1=can easily tolerate to 10=can't tolerate at all. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A negative change from Baseline indicated an improvement (less impact of tooth sensitivity on participant's everyday life).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Baseline (Day 0) | 5.66 (1.987) | 5.32 (1.939) | 4.77 (1.668) | 4.86 (1.552)
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 3 | -0.62 (1.208) | 0.04 (1.036) | -0.28 (0.841) | -0.21 (1.343)
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 14 | -1.37 (1.757) | -0.83 (1.947) | -1.00 (1.114) | -0.45 (1.703)
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 28 | -1.04 (1.791) | -0.93 (1.617) | -1.10 (1.373) | -0.81 (1.575)
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Q7 (On a scale of 1 to 10 how intense are the sensations?): Change from Baseline at Day 56 | -1.07 (1.850) | -1.39 (1.838) | -1.77 (1.431) | -0.86 (1.820)
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Baseline (Day 0) | 5.10 (2.540) | 4.97 (2.008) | 4.52 (2.111) | 4.41 (2.009)
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 3 | -0.21 (1.082) | -0.18 (1.335) | -0.34 (1.143) | 0.00 (1.491)
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 14 | -0.59 (2.206) | -0.76 (1.766) | -0.83 (1.085) | -0.21 (1.719)
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 28 | -0.48 (1.896) | -1.00 (1.390) | -0.83 (1.533) | -0.46 (1.529)
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Q8 (On a scale of 1 to 10 how bothered are you by any sensations?): Change from Baseline at Day 56 | -0.52 (1.883) | -1.06 (1.413) | -1.63 (1.351) | -0.57 (2.150)
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Baseline (Day 0) | 4.93 (2.563) | 4.39 (2.261) | 3.77 (2.202) | 3.83 (2.054)
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 3 | -0.14 (2.065) | 0.29 (1.150) | 0.17 (1.605) | 0.18 (2.178)
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 14 | -0.81 (2.058) | 0.24 (1.845) | -0.27 (1.143) | 0.48 (2.707)
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 28 | -0.76 (1.535) | -0.17 (1.913) | -0.47 (2.013) | -0.27 (2.201)
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Q9 (On a scale of 1 to 10 how well can you tolerate sensations?): Change from Baseline at Day 56 | -0.52 (2.148) | -0.10 (2.119) | -0.90 (2.155) | -0.29 (2.692)

19. Secondary Outcome: Change From Baseline in DHEQ Total Score (Section 2 Questions 1-15) at Days 3, 14, 28 and 56
Description: DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of 2 sections. Section 2 included 15 questions about the ways in which sensations in participant's teeth affected them in their daily life. Questions were grouped into the following domains: Restrictions(Q1-3), Adaptation(Q4-6), Social Impact(Q7-9), Emotional Impact(Q10-12), and Identity(Q13-15). All participants scored 15 questions using a 7-point scale, where 7=Strongly agree, 6=Agree, 5=Agree a little, 4=neither agree or disagree, 3=disagree a little, 2=disagree, and 1=strongly disagree. Total score was derived from the sum of scores in single domains and ranged from 15 to 105. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting Baseline value from value at each indicated timepoint. A negative change from Baseline indicated improvement (less impact of sensations on participant's daily life).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 67.41 (17.235) | 60.06 (18.703) | 57.19 (17.651) | 61.79 (19.580)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | 0.62 (7.370) | -1.71 (11.132) | -1.93 (3.283) | -0.71 (11.524)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | -0.48 (10.271) | -4.41 (12.701) | -6.00 (11.750) | -1.55 (11.624)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -1.80 (11.979) | -4.53 (14.176) | -7.63 (13.071) | -3.04 (13.250)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -2.38 (13.808) | -8.61 (16.508) | -10.67 (14.456) | -4.00 (13.411)

20. Secondary Outcome: Change From Baseline in DHEQ Restrictions Domain Score (Section 2 Questions 1 to 3) at Days 3, 14, 28 and 56
Description: DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of 2 sections. Restriction domain(Q1 to 3) of Section 2 consisted of following questions: Q1:Having sensation in my teeth takes a lot of the pleasure out of eating and drinking; Q2:It takes a long time to finish some foods and drinks because of sensations in my teeth; Q3:There have been times when I have had problems eating ice cream because of these sensations. All participants scored Q1 to 3 using a 7-point scale, where 7=Strongly agree, 6=Agree, 5=Agree a little, 4=neither agree or disagree, 3=disagree a little, 2=disagree, and 1=strongly disagree. Total score ranged from 3 to 21. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting Baseline value from value at each indicated timepoint. A negative change from Baseline indicated improvement(less impact of sensations on participant's daily life).
Time Frame: Baseline (Day 0), Days 3, 14, 28, 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 15.14 (3.916) | 13.32 (4.854) | 12.03 (4.505) | 13.72 (4.651)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | 0.10 (1.655) | -0.50 (2.963) | -0.21 (1.989) | 0.29 (3.029)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | -0.85 (3.110) | -1.52 (3.334) | -1.13 (3.148) | 0.03 (2.970)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -0.44 (3.809) | -1.13 (3.411) | -1.47 (3.148) | -1.04 (2.807)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -0.83 (3.174) | -1.90 (3.736) | -2.27 (3.877) | -0.50 (3.085)

21. Secondary Outcome: Change From Baseline in DHEQ Adaptation Domain Score (Section 2 Questions 4 to 6) at Days 3, 14, 28 and 56
Description: DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of 2 sections. Adaptation domain (Q4 to 6) of Section 2 consisted of following questions: Q4: I have to change the way I eat or drink certain things; Q5: I have to be careful how I breathe on a cold day; Q6: When eating some foods, I have made sure they don't touch certain teeth. All participants scored Q4 to 6 using a 7-point scale, where 7= Strongly agree, 6=Agree, 5=Agree a little, 4=neither agree or disagree, 3=disagree a little, 2=disagree, and 1=strongly disagree. Total score ranged from 3 to 21. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A negative change from Baseline indicated improvement (less impact of sensations on participant's daily life).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 14.55 (4.197) | 13.48 (4.335) | 13.26 (4.000) | 13.38 (4.135)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | 0.17 (2.054) | -0.93 (3.005) | -0.62 (1.720) | 0.00 (2.944)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | -0.07 (3.292) | -1.24 (3.313) | -2.30 (3.153) | -0.62 (3.570)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -0.64 (3.581) | -1.57 (4.360) | -2.10 (4.063) | -0.85 (3.068)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -0.79 (3.940) | -2.19 (4.629) | -3.33 (3.809) | -1.14 (3.638)

22. Secondary Outcome: Change From Baseline in DHEQ Social Impact Domain Score (Section 2 Questions 7 to 9) at Days 3, 14, 28 and 56
Description: DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of 2 sections. Social Impact domain(Q7 to 9) of Section 2 consisted of following questions: Q7:Because of sensations I take longer than others to finish meal; Q8:I have to be careful what I eat when I am with others because of sensation in my teeth; Q9:Going to dentist is hard for me because I know it is going to be painful as a result of sensations in my teeth. All participants scored Q7 to 9 using a 7-point scale, where 7=Strongly agree, 6=Agree, 5=Agree a little, 4=neither agree or disagree, 3=disagree a little, 2=disagree, and 1=strongly disagree. Total score ranged from 3 to 21. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting Baseline value from value at each indicated timepoint. A negative change from Baseline indicated improvement(less impact of sensations on participant's daily life).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 11.38 (4.354) | 10.26 (4.099) | 9.74 (3.803) | 10.59 (4.961)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | 0.38 (2.007) | -0.04 (2.457) | -0.38 (2.060) | -0.32 (2.420)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | 0.67 (2.094) | -0.62 (3.075) | -0.57 (2.473) | -0.03 (2.368)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -0.04 (2.525) | -0.17 (3.705) | -1.00 (2.792) | -0.38 (3.579)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | 0.38 (3.156) | -1.00 (3.733) | -1.43 (2.873) | -0.57 (2.974)

23. Secondary Outcome: Change From Baseline in DHEQ Emotional Impact Domain Score (Section 2 Questions 10 to 12) at Days 3, 14, 28 and 56
Description: DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of 2 sections. Emotional Impact domain (Q10 to 12) of Section 2 consisted of following questions: Q10: I have been anxious that something I eat, or drink might cause sensations in my teeth; Q11: The sensations in my teeth have been irritating; Q12: The sensations in my teeth have been annoying. All participants scored Q10 to 12 using a 7-point scale, where 7= Strongly agree, 6=Agree, 5=Agree a little, 4=neither agree or disagree, 3=disagree a little, 2=disagree, and 1=strongly disagree. Total score ranged from 3 to 21. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A negative change from Baseline indicated improvement (less impact of sensations on participant's daily life).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 14.93 (3.474) | 13.10 (4.452) | 12.45 (3.695) | 13.38 (4.716)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | 0.17 (3.402) | -0.04 (3.156) | -0.31 (2.189) | 0.25 (4.151)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | -0.48 (3.081) | -0.69 (3.444) | -1.20 (3.284) | -0.07 (3.990)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -0.64 (2.856) | -0.63 (3.378) | -1.70 (3.743) | -0.38 (5.146)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -0.48 (3.631) | -1.81 (4.293) | -2.77 (3.892) | -0.57 (4.367)

24. Secondary Outcome: Change From Baseline in DHEQ Identity Domain Score (Section 2 Questions 13 to 15) at Days 3, 14, 28 and 56
Description: DHEQ was a validated, condition-specific measure of the impacts of tooth sensitivity on everyday life. It consisted of 2 sections. Identity domain (Q13 to 15) of Section 2 consisted of following questions: Q13: Having these sensations in my teeth makes me feel old; Q14: Having these sensations in my teeth makes me feel damaged; Q15: Having these sensations in my teeth makes me feel as though I am unhealthy. All participants scored Q13 to 15 using a 7-point scale, where 7= Strongly agree, 6=Agree, 5=Agree a little, 4=neither agree or disagree, 3=disagree a little, 2=disagree, and 1=strongly disagree. Total score ranged from 3 to 21. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A negative change from Baseline indicated improvement (less impact of sensations on participant's daily life).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 11.41 (5.124) | 9.90 (4.392) | 9.71 (4.451) | 10.72 (4.963)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | -0.21 (2.704) | -0.21 (2.794) | -0.41 (1.862) | -0.93 (2.595)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | 0.26 (3.265) | -0.34 (3.528) | -0.80 (2.280) | -0.86 (3.193)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -0.04 (2.746) | -1.03 (3.409) | -1.37 (2.220) | -0.38 (2.886)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -0.66 (3.330) | -1.71 (3.349) | -0.87 (3.277) | -1.21 (3.190)

25. Secondary Outcome: Mean Numeric Rating Scale (NRS) Score at Baseline, Days 3, 14, 28 and 56
Description: The NRS was a segmented numeric version of the visual analog scale (VAS) in which a participant selected a number from 0 to 10 that best reflected the intensity of the discomfort caused by sensitivity in their teeth, where 0=no discomfort and 10=worst discomfort imaginable. Lower score indicated less discomfort caused by the sensitivity.
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 5.3 (2.55) | 5.1 (1.98) | 4.6 (1.69) | 4.3 (2.24)
  Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Day 3 | 4.9 (2.50) | 5.0 (2.05) | 4.2 (1.68) | 4.5 (1.80)
  Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Day 14 | 4.4 (2.41) | 4.5 (1.92) | 3.5 (1.50) | 4.3 (2.04)
  Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Day 28 | 4.6 (2.33) | 4.0 (2.19) | 3.2 (1.95) | 4.2 (1.56)
  Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Day 56 | 4.4 (2.29) | 3.6 (2.23) | 2.7 (1.80) | 3.8 (2.18)

26. Secondary Outcome: Change From Baseline in Mean NRS Score at Days 3, 14, 28 and 56
Description: The NRS was a segmented numeric version of the VAS in which a participant selected a number from 0 to 10 that best reflected the intensity of the discomfort caused by sensitivity in their teeth, where 0=no discomfort and 10=worst discomfort imaginable. Lower score indicated less discomfort caused by the sensitivity. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. A negative change from Baseline indicated improvement (reduction in discomfort caused by sensitivity).
Time Frame: Baseline (Day 0), Days 3, 14, 28 and 56
Population: The mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
Number analyzed (Participants) | 29 | 31 | 31 | 29
score on a scale
  Baseline (Day 0) | 5.3 (2.55) | 5.1 (1.98) | 4.6 (1.69) | 4.3 (2.24)
  Change from Baseline at Day 3: number analyzed (Participants) | 29 | 28 | 29 | 28
  Change from Baseline at Day 3 | -0.5 (1.09) | -0.1 (1.36) | -0.4 (1.35) | 0.2 (1.85)
  Change from Baseline at Day 14: number analyzed (Participants) | 27 | 29 | 30 | 29
  Change from Baseline at Day 14 | -0.9 (1.96) | -0.7 (1.99) | -1.1 (1.78) | -0.0 (2.38)
  Change from Baseline at Day 28: number analyzed (Participants) | 25 | 30 | 30 | 26
  Change from Baseline at Day 28 | -0.9 (1.67) | -1.1 (2.09) | -1.4 (1.91) | -0.3 (2.23)
  Change from Baseline at Day 56: number analyzed (Participants) | 29 | 31 | 30 | 28
  Change from Baseline at Day 56 | -0.9 (2.09) | -1.5 (2.32) | -1.9 (1.54) | -0.6 (2.26)

ADVERSE EVENTS:
Time Frame: Baseline up to 5 days after last use of study product (up to approximately 61 days)
Description: Adverse events (AEs) were to be collected for Safety population and were defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study product including any acclimatisation, washout or leadin product (or medical device). A Serious AE (SAE) was a particular category of an AE where the adverse outcome was serious. However, no deaths, AEs or SAEs were reported.
Arm/Group | Test Product | Comparator 1 | Comparator 2 | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31 | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT05243745/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT05243745/SAP_001.pdf